CLINICAL TRIAL: NCT04447846
Title: Novel Cognitive Treatment Targets for Epidiolex in Sturge- Weber Syndrome: A Phase II Trial
Brief Title: Novel Cognitive Treatment Targets for Epidiolex in Sturge- Weber Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anne Comi, MD (Other)
Collaborators: Jazz Pharmaceuticals (Industry); Faneca 66 Foundation (Other)
Responsible Party: Sponsor-Investigator, Anne Comi, MD, Principal Investigator, Director Sturge-Weber Center, Kennedy Krieger Institute, Professor Johns Hopkins University School of Medicine, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Organization: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00204427
Record Dates: First submitted 2019-10-10; First posted 2020-06-25 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Sturge-Weber Syndrome
Keywords: Sturge-Weber Syndrome; SWS; Cognitive impairments
MeSH Terms: conditions — Sturge-Weber Syndrome; Cognitive Dysfunction | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cannabidiol/ Epidiolex (Experimental): All subjects will receive the experimental Epidiolex (cannabidiol) oral solution to be taken at home twice a day, and will be treated on an outpatient basis. The drug will be taken for 24 weeks unless the subject chooses to participate in the extension phase of the study, in which case the subject will continue to receive the drug for one additional year or until the drug is approved for clinical use for the treatment of cognitive impairments in patients with Sturge-Weber syndrome.
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Initiation of treatment will begin with 5 mg/kg/day given in two divided doses. The dose will be increased by 5 mg/kg/day after seven days and then by 5 mg/kg/day every seven days up to a maximum dose of 20 mg/kg/day given.
  Other Names: Epidiolex; CBD

SUMMARY:
The purpose of this study is to better understand the utility of cannabidiol (CBD/ Epidiolex) for improving the treatment of cognitive impairments in Sturge-Weber syndrome (SWS).

DETAILED DESCRIPTION:
The investigators hope to gain an understanding of the utility of pharmaceutical grade CBD used for the treatment of cognitive impairments in SWS in this open-label study. Anecdotal evidence from a phase I trial investigating the use of CBD for medically refractory seizures suggests CBD may also have a beneficial effect on cognition, mood, and behavior. The investigators hypothesize that CBD/ Epidiolex will improve SWS brain function resulting in improved cognitive function, social interactions, mood, motor function and behavior, as well as reduced migraines. This is an open-label prospective oral drug trial of Epidiolex in 10 subjects. Assessments will be done at baseline and repeated after 6 months on study drug.

ELIGIBILITY:
Inclusion Criteria: Participants with Sturge-Weber syndrome brain involvement as defined on neuroimaging (n=10 subjects, male and female, ages 3 to 50 years of age) and the following:

* Cognitive impairment defined as a cognitive neuroscore greater than or equal to 2 at screening.
* Anti-epileptic, mood or behavioral drugs (if on) at stable doses for a minimum of 4 weeks prior to enrollment.
* If present, VNS must be on stable setting for a minimum of 3 months prior to enrollment.
* If on ketogenic or Atkins diet, must be on stable ratio for a minimum of 3 months prior to enrollment.
* Previous subjects who fail at any point to meet continuation criteria and withdraw early may be considered for re-enrollment under new subject ID as long as the above inclusion criteria are met. The determination of whether to re-enroll will be made by the PI and sponsor on a case-by-case basis. Re-enrollment can occur no earlier than 4 weeks after the final, post-weaning follow-up visit under the old subject ID.
* Written informed consent obtained from the patient or the patient's legal representative must be obtained prior to beginning treatment.

Exclusion Criteria:

* Patients with any severe and/or uncontrolled medical conditions at randomization such as:

  1. Liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis (i.e. quantifiable HBV-DNA and/or positive HbsAg, quantifiable HCV-RNA)
  2. Uncontrolled diabetes as defined by fasting serum glucose greater than 1.5
  3. Active (acute or chronic) or uncontrolled severe infections
  4. Active, bleeding diathesis
* Patients who have a major surgery or significant traumatic injury within 4 weeks of study entry, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia), or patients that may require major surgery during the course of the study.
* Patients who start or discontinue a seizure, mood or behavioral medication in the 4 weeks leading up to screening.
* Prior treatment with any investigational drug or use of any other cannabis product within the preceding 4 weeks prior to study entry.
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study. This includes those in foster care, or those unable to keep follow-up appointments, maintain close contact with the Principal Investigator, or complete all necessary studies to maintain safety.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of the female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2022-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Comi, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

REFERENCES:
- See also: Hunter Nelson Sturge-Weber Center Website — https://www.kennedykrieger.org/patient-care/centers-and-programs/sturge-weber-syndrome-center

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After consent, subject 10 was not enrolled as they did not meet the inclusion criteria of remaining at a stable does of anti-epileptic drugs 4 weeks prior to enrollment.
Period: Overall Study
Arm/Group | Cannabidiol/ Epidiolex
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrew due to moderate side effects (fatigue) | 1

BASELINE CHARACTERISTICS:
Groups:
- Cannabidiol: Subjects took oral cannabidiol for 6 months (doses ranged from 5 mg/kg/day to 20 mg/kg/day). Neuropsychological, psychiatrics and motor assessments were administered at baseline and six months follow-up.
Arm/Group | Cannabidiol
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.83 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 6
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10
Brain Involvement [Count of Participants; unit: Participants]
  Right-Sided Brain Involvement | 6
  Left-Sided Brain Involvement | 2
  Bilateral Brain Involvement | 2
Skin Involvement [Count of Participants; unit: Participants]
  Right-Sided Skin Involvement | 4
  Left-Sided Skin Involvement | 2
  Bilateral Skin Involvement | 4
Eye Involvement [Count of Participants; unit: Participants]
  Right-Sided Eye Involvement | 4
  Left-Sided Eye Involvement | 2
  Bilateral Eye Involvement | 1
  No Eye Involvement | 3

OUTCOME MEASURES:

1. Primary Outcome: List Sorting Working Memory Test
Description: Data on cognitive function was collected using the List Sorting Working Memory Test from the NIH Toolbox. Data was collected on working memory performance, which was transformed into a t-score from 0 to 100 where a higher t-score indicates better performance. T-score of 50 indicates the population mean with a standard deviation of 10. Data was collected at baseline and after 6 months on study drug.
Time Frame: Baseline, Follow-up (6 months)
Population: Subject 1 was unable to complete this assessment due to lack of understanding of the instructions. Subject 10 was unable to complete this assessment due to a system error, where the fully adjusted score was not obtained. Subject 9 was withdrawn prior to the 6 month follow-up visit due to a persistent side effect and was not included in analysis.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 7
T-score
  Baseline List Sorting Working Memory Fully Adjusted Score | 37.14 (10.92)
  Follow-Up List Sorting Working Memory Fully Adjusted Score | 39.14 (13.78)

2. Secondary Outcome: Picture Vocabulary Test
Description: Data on cognitive function was collected using the Picture Vocabulary subtest from the NIH Toolbox. Single words are presented via an audio file, paired simultaneously with 4 screen images of objects, actions, and/or depictions of concepts. The task is to pick the picture that matches the spoken word. Performance on the task was transformed into a t-score from 0 to 100 where a higher t-score indicates better performance. T-score of 50 indicates the population mean with a standard deviation of 10. Data was collected at baseline and after 6 months on study drug.
Time Frame: Baseline, Follow-up (6 months)
Population: Subject 10 did not complete this assessment due to a technical issue where the fully adjusted score was not calculated. Subject 9 was withdrawn from the study prior to the 6 month follow-up visit due to a persistent side effect and was not included in analysis.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 8
T-score
  Baseline Mean of the Fully Adjusted Picture Vocabulary Score | 42.88 (8.86)
  Follow-up Mean of the Fully Adjusted Picture Vocabulary Score | 42.38 (9.43)

3. Secondary Outcome: Seizure Frequency
Description: Change in seizure frequency by seizure score at pre-treatment baseline and after six months. The seizure score is taken from the Sturge-Weber Neuroscore on a scale of 0 to 4 where 0=none, 1=1+. but controlled, 2=Breakthrough, 3=monthly, 4=Weekly+. Higher scores indicate worse outcome.
Time Frame: Baseline, Follow-up (6 months)
Population: Subject 9 was withdrawn prior to the 6 month follow-up visit due to a persistent side effect and was not included in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 9
score on a scale
  Baseline Seizure Score from Sturge-Weber Neuroscore | 1.11 (0.33)
  Follow-up Seizure Score from Sturge-Weber Neuroscore | 1.00 (0.00)

4. Secondary Outcome: Migraine Severity
Description: Data on migraine severity will be collected using patient responses to questions on a standard six-point scale. Data will be collected on the frequency of an event (e.g. feelings of frustration, performance of daily activities) which will be transformed into a score from 0 to 100 where higher scores indicate a less migraine severity and better outcomes. Data will be collected at baseline and after 6 months on study drug.
Time Frame: Baseline, Follow-up (6 months)
Population: Subject 7 misplaced this questionnaire and was not included in analysis. Subject 9 was withdrawn prior to the 6 month follow-up visit due to a persistent side effect and was not included in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 8
score on a scale
  Baseline Mean Migraine-Quality of Life Score | 96.83 (7.62)
  Follow-up Mean Migraine-Quality of Life Score | 97.50 (4.69)

5. Secondary Outcome: Modified House Classification Scores
Description: Data on motor function was collected using a Modified House Classification. Data was collected on the ability to complete a task with the subject's non-dominant hand which was transformed into a score from 1 to 8 and 0 to 32 where higher scores indicate better motor function. Data was collected at baseline and after 6 months on study drug.
Time Frame: Baseline, Follow-up (6 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 9
score on a scale
  Baseline Mean Highest Category in Which All Items were Successfully Completed | 5.11 (0.93)
  Follow-up Mean Highest Category in Which All Items were Successfully Completed | 5.44 (1.33)
  Baseline Mean Total Number of Items Successfully Completed | 26.67 (4.12)
  Follow-up Mean Total Number of Items Successfully Completed | 27.44 (4.75)

6. Secondary Outcome: Erhardt Developmental Prehension Assessment Scores
Description: Data on motor function was collected using the Erhardt Developmental Prehension assessment. Data was collected on the ability to complete a task with each hand, which was scored as age equivalence of task performance (in months). Higher scores indicate better motor function. Data was collected at baseline and after 6 months on study drug.
Time Frame: Baseline, Follow-up (6 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 9
Months
  Baseline Mean Dominant Hand Total Score | 54.22 (2.64)
  Follow-up Mean Dominant Hand Total Score | 53.56 (4.04)
  Baseline Mean Non-Dominant Hand Total Score | 51.22 (9.48)
  Follow-up Mean Non-Dominant Hand Total Score | 53.78 (4.15)

7. Secondary Outcome: Pediatric Evaluation of Disability Inventory Computer Adapted Test
Description: Data on motor function was collected using the Pediatric Evaluation of Disability Inventory Computer Adapted Test. Data was collected on the subject's ability to complete tasks involved in daily activities, mobility, and social/ cognitive activities. The data was transformed into scaled scores ranging from 20 to 80, where higher scores indicate better motor function. Data was collected at baseline and after 6 months on study drug.
Time Frame: Baseline, Follow-up (6 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 9
score on a scale
  Baseline Mean Score for Daily Activities | 58.67 (7.76)
  Follow-up Mean Score for Daily Activities | 60.00 (6.50)
  Baseline Mean Score for Mobility | 67.11 (4.76)
  Follow-Up Mean Score for Mobility | 68.56 (4.07)
  Baseline Mean Score for Responsibility | 52.44 (11.67)
  Follow-Up Mean Score for Responsibility | 53.89 (11.10)
  Baseline Mean Score for Social Cognitive | 66.89 (5.35)
  Follow-up Mean Score for Social Cognitive | 67.22 (4.63)

8. Secondary Outcome: ABILHAND Questionnaire
Description: Data on motor function was collected using the ABILHAND questionnaire, a measure of manual ability for adults with upper limb impairments. Data was collected on the subject's ability to complete daily activities that involve the upper limbs. Score was collected as a patient measure with scores ranging from -10 to 10. Higher scores indicate better motor function. Data was collected at baseline and after 6 months on study drug.
Time Frame: Baseline, Follow-up (6 months)
Population: Subject 7 misplaced this questionnaire and was not included in analysis. Subject 9 was withdrawn prior to the 6 month follow-up visit due to persistent side effect and was not included in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 8
score on a scale
  Baseline Mean of the ABILHAND | 1.81 (1.98)
  Follow-up Mean of the ABILHAND | 2.88 (1.39)

9. Secondary Outcome: Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V) or Wechsler Adult Intelligence Scale (WAIS-IV)
Description: Data on cognitive function was collected using selected subtests, from either the Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V) or the Wechsler Adult Intelligence Scale (WAIS-IV). For the WISC-V and WAIS-IV subtests selected, scaled scores were derived from the normative data which account for age and demographic information. The selected WISC-V/WAIS-IV subtests were as follows: Digit Span, Symbol Search, Coding and Processing Speed; the first three subtests were scored from 0-10, the fourth subtest from 0-100, and for all subtests higher score is better. The selected subtests, from the WISC-V and the WAIS-IV, were combined to increase statistical power.
  Statistically rare changes in individual test scores were determined using a reliable change index methodology based upon normative information for these assessments.
Time Frame: Baseline, Follow-up (6 months)
Population: Subjects 1 and 10 did not complete this questionnaire as they were too young. Subject 9 was withdrawn prior to the 6 month follow-up visit due to a persistent side effect and was not included in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 7
score on a scale
  Baseline Mean Digit Span Score | 5.71 (2.81)
  Follow-up Mean Digit Span Score | 6.43 (2.07)
  Baseline Mean Symbol Search Score | 6.00 (2.71)
  Follow-up Mean Symbol Search Score | 5.57 (2.07)
  Baseline Mean Coding Score | 5.57 (2.88)
  Follow-up Mean Coding Score | 4.71 (2.22)
  Baseline Mean Processing Speed Score | 77.14 (13.93)
  Follow-up Mean Processing Speed Score | 73.43 (11.19)

10. Secondary Outcome: Pediatric Neurological Quality of Life (Neuro-QoL)
Description: Data on cognitive function was collected using Neurological Quality of Life scales from the NIH Toolbox. Data on frequency of an event (e.g. forgetting schoolwork) was collected and transformed into a t-score from 0 to 100 where higher t-scores indicate worse anger, worse anxiety, worse pain, better social relationships, worse stigma, worse depression, better cognitive function, and worse fatigue. T-score of 50 indicates the population mean with a standard deviation of 10. Data was collected at baseline and 6 months on study drug.
Time Frame: Baseline, Follow-up (6 months)
Population: Subjects below the age of 18 completed the pediatric version of this questionnaire and were included in analysis.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 6
T-score
  Baseline Mean Pediatric Score for Anger | 53.02 (3.09)
  Follow-up Mean Pediatric Score for Anger | 49.67 (7.00)
  Baseline Mean Pediatric Score for Anxiety | 45.20 (5.79)
  Follow-up Mean Pediatric Score for Anxiety | 41.07 (5.74)
  Baseline Mean Pediatric Score for Pain | 40.20 (4.16)
  Follow-up Mean Pediatric Score for Pain | 43.50 (5.89)
  Baseline Mean Pediatric Score for Social Relations | 43.28 (15.10)
  Follow-up Mean Pediatric Score for Social Relations | 54.33 (6.96)
  Baseline Mean Pediatric Score for Stigma | 42.45 (6.42)
  Follow-up Mean Pediatric Score for Stigma | 44.52 (4.88)
  Baseline Mean Pediatric Score for Depression | 44.07 (6.29)
  Follow-up Mean Pediatric Score for Depression | 44.62 (8.58)
  Baseline Mean Pediatric Score for Cognitive Function | 49.27 (3.36)
  Follow-up Mean Pediatric Score for Cognitive Function | 51.33 (6.44)
  Baseline Mean Pediatric Score for Fatigue | 46.38 (9.44)
  Follow-up Mean Pediatric Score for Fatigue | 45.97 (8.14)

11. Secondary Outcome: Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2)
Description: Data on executive function was collected using the Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2). Data on the frequency of an event (e.g. becomes upset too easily) was collected and transformed into a t-score. The following BRIEF-2 subtests were evaluated: Behavioral Regulation Index, Emotional Regulation Index, Cognitive Regulation Index, and Global Executive Composite. For each BRIEF-2 subtest, t-scores range from 0 to 100; a score of 50 indicates the population mean with a standard deviation of 10. For all BASC-3 subtests, higher scores are worse outcome.
Time Frame: Baseline, Follow-up (6 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 9
T-score
  Baseline Mean for Behavioral Regulation Index | 55.11 (11.66)
  Follow-Up Mean for Behavioral Regulation Index | 52.44 (13.60)
  Baseline Mean for Emotional Regulation Index | 60.22 (10.24)
  Follow-up Mean for Emotional Regulation Index | 51.22 (12.29)
  Baseline Mean for Cognitive Regulation Index | 54.11 (7.06)
  Follow-up Mean for Cognitive Regulation Index | 54.22 (10.59)
  Baseline Mean for Global Executive Composite | 56.78 (8.17)
  Follow-up Mean for Global Executive Composite | 53.33 (11.57)

12. Secondary Outcome: Social Responsiveness Scale, Second Edition (SRS-2)
Description: Data on social function was collected using the Social Responsiveness Scale-Second Edition (SRS-2). Data on a child's ability to engage in emotionally appropriate reciprocal social interactions in naturalistic settings was collected and transformed into a t-score from 0 to 100 where higher scores indicate greater impairment in social function. T-score of 50 indicates the population mean with a standard deviation of 10. Data was collected at baseline and 6 months on study drug.
Time Frame: Baseline, Follow-up (6 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 9
T-score
  Baseline Mean Total Score | 54.22 (7.71)
  Follow-up Mean Total Score | 49.22 (7.09)

13. Secondary Outcome: Behavioral Assessment System for Children, Third Edition (BASC-3)
Description: Data on behavioral function was collected using the Behavioral Assessment System for Children, Third Edition (BASC-3). Data on the frequency of a behavior (e.g. avoids eye contact) was collected and transformed into a t-score. Subscales for the BASC-3 scored were: External Problems Composite, the Internal Problems Composite, the Behavioral Symptoms Index, and the Adaptive Skills Composite. For the first three subscales, lower t-score indicates better outcome; for the fourth, a lower t-score indicates worse outcome. T-scores for all the BASC-3 subscales range from 0 to 100, and a t-score of 50 indicates the population mean with a standard deviation of 10.
Time Frame: Baseline, Follow-up (6 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 9
T-score
  Baseline Mean External Problems Composite | 51.22 (6.10)
  Follow-up Mean External Problems Composite | 50.11 (6.31)
  Baseline Mean Internal Problems Composite | 52.22 (5.81)
  Follow-Up Mean Internal Problems Composite | 46.22 (7.17)
  Baseline Mean Behavioral Symptoms Index | 54.22 (4.21)
  Follow-up Mean Behavioral Symptoms Index | 50.11 (8.19)
  Baseline Mean Adaptive Skills Composite | 45.00 (8.29)
  Follow-Up Mean Adaptive Skills Composite | 48.44 (7.63)

14. Secondary Outcome: Screen for Child Anxiety Related Disorders (SCARED)
Description: Data on anxiety was collected using the Screen for Child Anxiety Related Disorders (SCARED). Data on the truthfulness of a statement (e.g. I am nervous) was collected and transformed into a score from 0 to 82 where higher scores indicate greater anxiety. Data was collected at baseline and 6 months on study drug.
Time Frame: Baseline, Follow-up (6 months)
Population: Subject 7 misplaced this assessment and was not included in analysis. Subject 9 was withdrawn from the study prior to the 6 month follow-up visit due to a persistent side effect and was not included in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 8
score on a scale
  Baseline Mean of Total Score | 14.86 (14.49)
  Follow-up Mean of Total Score | 11.57 (11.16)

15. Secondary Outcome: Quality of Life in Childhood Epilepsy Questionnaire (QOLCE-55)
Description: Data on quality of life was collected using the Quality of Life in Childhood Epilepsy Questionnaire (QOLCE-55). Data on the frequency of an event (e.g. had trouble concentrating on a task) was collected and transformed into a score from 0 to 100 where higher scores reflect better quality of life. Data was collected at baseline and 6 months on study drug.
Time Frame: Baseline, Follow-up (6 months)
Population: Subject 7 misplaced this assessment and was not included in analysis. Subject 9 was withdrawn prior to the 6 month follow-up appointment due to a persistent side effect and was not included in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 8
score on a scale
  Baseline Mean Total Score | 61.17 (18.14)
  Follow-up Mean Total Score | 71.39 (10.75)

16. Secondary Outcome: Safety of Epidiolex
Description: Safety of Epidiolex was measured by the number of adverse events and serious adverse events that result from study drug.
Time Frame: Baseline, Follow-up (6 months)
Measure: Number; unit: Events
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 10
Events
  Number of Adverse Events that Resulted from the Study Drug | 24
  Number of Serious Adverse Events that Resulted from the Study Drug | 0

17. Secondary Outcome: Neuroscore
Description: Data on neurological function was collected using the Neuroscore. Data on frequency of seizures, extent of hemiparesis, assessment of visual field cut, and degree of cognitive functioning was transformed into a score from 0 to 15 where higher scores indicate worse neurologic function. Data was collected at baseline and 6 months on study drug.
Time Frame: Baseline, Follow-up (6 months)
Population: Subject 9 was withdrawn prior to the 6 month follow-up visit and not included in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 9
score on a scale
  Baseline Mean Seizure Score | 1.11 (0.33)
  Follow-Up Mean Seizure Score | 1.00 (0.00)
  Baseline Mean Hemiparesis Score | 1.44 (1.13)
  Follow-Up Mean Hemiparesis Score | 1.00 (0.87)
  Baseline Mean Visual Field Cut Score | 0.11 (0.33)
  Follow-Up Mean Visual Field Cut Score | 0.00 (0.00)
  Baseline Mean Cognitive Function Score | 2.33 (0.50)
  Follow-up Mean Cognitive Function Score | 1.44 (0.53)
  Baseline Mean Composite Score | 5.00 (1.32)
  Follow-up Mean Composite Score | 3.44 (0.88)

18. Secondary Outcome: Port-wine Birthmark Score
Description: Data on facial port-wine birthmarks was collected using the Port-wine Birthmark Score. Data on percent of face covered, thickness of birthmark, and darkness of birthmark color was collected and transformed into a score from 0 to 43 where higher scores indicate greater severity and greater surface area involved. Data was collected at baseline and 6 months on study drug.
Time Frame: Baseline, Follow-up (6 months)
Population: Subject 9 was withdrawn prior to the 6 month follow-up appointment and was not included in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 9
score on a scale
  Baseline Mean Total Score | 8.56 (3.09)
  Follow-up Mean Total Score | 8.11 (3.18)

19. Secondary Outcome: Adult Neurological Quality of Life (Neuro-QoL)
Description: Data on cognitive function was collected using Neurological Quality of Life scales from the NIH Toolbox. Data on frequency of an event was collected and transformed into a t-score from 0 to 100. Higher t-scores indicate better communication, better ability to participate in social activity, worse anxiety, worse depression, worse emotional and behavioral dyscontrol, worse fatigue, better positive affect, worse sleep disturbance, better lower and upper extremity functions, worse stigma, better satisfaction with social roles, and better cognitive function. T-score of 50 indicates the population mean with a standard deviation of 10. Data was collected at baseline and 6 months on study drug.
Time Frame: Baseline, Follow-up (6 months)
Population: Subjects above the age of 18 completed the pediatric version of this questionnaire and were included in analysis.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cannabidiol/ Epidiolex
Number analyzed (Participants) | 3
T-score
  Baseline Mean Adult Score for Anxiety | 46.77 (13.33)
  Follow-Up Mean Adult Score for Anxiety | 46.87 (6.45)
  Baseline Mean Adult Score for Depression | 42.70 (10.05)
  Follow-Up Mean Adult Score for Depression | 44.23 (9.53)
  Baseline Mean Adult Score for Fatigue | 45.23 (9.53)
  Follow-Up Mean Adult Score for Fatigue | 42.80 (4.60)
  Baseline Mean Adult Score for Upper Extremity Function | 48.97 (8.37)
  Follow-Up Mean Adult Score for Upper Extremity Function | 53.80 (0.00)
  Baseline Mean Adult Score for Lower Extremity Function | 58.60 (0.00)
  Follow-Up Mean Adult Score for Lower Extremity Function | 58.60 (0.00)
  Baseline Mean Adult Score for Cognitive Function | 47.03 (15.52)
  Follow-Up Mean Adult Score for Cognitive Function | 46.73 (5.01)
  Baseline Mean Adult Score for Emotional and Behavioral Dyscontrol | 51.10 (14.97)
  Follow-Up Mean Adult Score for Emotional and Behavioral Dyscontrol | 41.37 (9.98)
  Baseline Mean Adult Score for Well-being | 54.30 (4.91)
  Follow-Up Mean Adult Score for Well-being | 55.70 (6.59)
  Baseline Mean Adult Score for Sleep Disturbances | 47.03 (7.49)
  Follow-Up Mean Adult Score for Sleep Disturbances | 43.93 (4.90)
  Baseline Mean Adult Score for Participation in Social Activities | 53.00 (7.41)
  Follow-Up Mean Adult Score for Participation in Social Activities | 51.03 (8.01)
  Baseline Mean Adult Score for Satisfaction in Social Activities | 47.70 (3.28)
  Follow-Up Mean Adult Score for Satisfaction in Social Activities | 49.23 (2.54)
  Baseline Mean Adult Score for Stigma | 53.90 (8.80)
  Follow-Up Mean Adult Score for Stigma | 56.47 (6.25)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Serious adverse events include those events that: result in death; are life-threatening; require hospitalization or prolongation of existing hospitalization; create persistent, significant disability, or birth defects.
  Expected adverse events are those that are identified in the research protocol as having been previously associated with participation in the study. All reported adverse events will be classified using the Common Terminology Criteria for Adverse Events Version 4.0.
Arm/Group | Cannabidiol/ Epidiolex
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cannabidiol/ Epidiolex (N=10)
Darkening of port-wine birthmark (Skin and subcutaneous tissue disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Ear and labyrinth disorders) | 2 (3)
Fatigue (Metabolism and nutrition disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (3)
Increased alanine aminotransferase (Hepatobiliary disorders) | 2 (2)
Increased aspartate aminotransferase (Hepatobiliary disorders) | 2 (2)
Irritable mood (Psychiatric disorders) | 1 (1)
Jitteriness (Psychiatric disorders) | 1 (1)
Mouth sores (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)

LIMITATIONS AND CAVEATS:
Due to the COVID-19 , visits transitioned from an in-person setting to a remote setting. Four subjects had baseline testing conducted in person and follow-up virtually, and 5 subjects had both baseline and follow-up testing virtually. The differences in testing environment and the context of the pandemic may have affected results. Also, due to variability in subject age and the small number of subjects, some participants were outside of assessment age norms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT04447846/Prot_SAP_000.pdf